CLINICAL TRIAL: NCT05822973
Title: Absorbable Versus Nonabsorbable Sutures for the Treatment of Knee Arthroscopy: A Prospective Comparison of Patient Outcomes and Satisfaction
Brief Title: Sutures for Treatment of Knee Arthroscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rothman Institute Orthopaedics (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KFRE18D.721
Record Dates: First submitted 2023-04-10; First posted 2023-04-21 (Actual); Last update posted 2023-04-21 (Actual); Status verified 2023-04

CONDITIONS: Knee Arthroscopy; Suture

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- would closure using absorbable sutures (Active Comparator): patients randomized into the absorbable suture group will have their incisions closed with 3.0 monocryl sutures
  Interventions: Device: 3.0 monocryl suture
- would closure using non-absorbable sutures (Active Comparator): Patients randomized into the nonabsorbable suture group will have their incisions closed with either a 3.0 nylon suture
  Interventions: Device: 3.0 nylon suture

INTERVENTIONS:
Device: 3.0 monocryl suture — incision will be closed with absorbable suture
  Arms: would closure using absorbable sutures
Device: 3.0 nylon suture — incision will be closed with non-absorbable suture
  Arms: would closure using non-absorbable sutures

SUMMARY:
For a knee arthroscopy, two small incisions are made at the level of the joint line on each side of the patellar tendon. Closure of surgical incisions consists of using either nonabsorbable or absorbable sutures. Some surgeons prefer using nonabsorbable sutures due to it being easier to tie, these sutures are less likely to break prematurely, and that they elicit a minimal inflammatory response. On the other hand, some surgeons prefer using absorbable sutures due to the time savings of not having to remove the sutures at a later date and that these sutures decrease patient anxiety and discomfort. The purpose of this study is to prospectively investigate and compare patient's pain, swelling and cosmesis following knee arthroscopy surgery between patients who had their arthroscopy portals closed using resorbable sutures vs. patients who had their portals closed using nonabsorbable sutures.

ELIGIBILITY:
Inclusion Criteria:

* Patients ages 18 and older undergoing primary knee arthroscopy for diagnostic arthroscopy, removal of a loose body, chondroplasty, or a partial meniscectomy will be included in this analysis

Exclusion Criteria:

* Patients undergoing revision knee arthroscopy as well as patients undergoing ACL reconstruction or meniscal repair surgery will be excluded from this analysis.
* Patients under the age of 18 will be excluded as well.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 274 (Actual)
Dates: Start 2018-11-18 (Actual); Primary Completion 2023-04-09 (Actual); Study Completion 2023-04-09 (Actual)

PRIMARY OUTCOMES:
Postoperative Pain Leveles | 3 months
  Pain levels will be recorded through the Visual Analogue Scale (VAS)
Patient Satisfaction | 3 months
  Satisfaction will be measures with customized questions regarding the overall satisfaction of their incision (on a scale of 0 to 10), satisfaction of the suture removal process, complications and swelling

CONTACTS AND LOCATIONS:
Locations (1):
- Rothman Orthopaedic Institute, Philadelphia, Pennsylvania, United States